CLINICAL TRIAL: NCT01546428
Title: A Phase I Study of INC280 in Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X1101
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-06

CONDITIONS: Advanced Solid Tumor
Keywords: c-MET; Advanced solid tumor
MeSH Terms: interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INC280 (Experimental)
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280

SUMMARY:
INC280 will be administered to Japanese patients with advanced soid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists. The trial will assess the safety and tolerability and determine the maximum tolerated dose (MTD) on INC280

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors that are refractory to currently available therapies or for which no effective treatment is available.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Good organ (hepatic, kidney, BM) function at screening/baseline visit.

Exclusion criteria:

* Symptomatic CNS metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of INC280.
* Undergone a bone marrow or solid organ transplant.
* Women who are pregnant or breast feeding.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) in the dose escalation part | 4 weeks
  Incidence and frequency of DLT during the first cycle of INC280 treatment in the dose escalation part according to the CTCAE.

SECONDARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events, changes in laboratory values | 4 months
  Incidence and severity of adverse events and serious adverse events, changes in laboratory values will be measured during the treatment.
Plasma concentration of INC280 and derived PK parameters of INC280 such as Tmax, AUC and T1/2 | 1 month
  Plasma concentration of INC280 and derived PK parameters of INC280 will be measured with serial plasma samples during treatment for first months.
Preliminary tumor responses according to RECIST 1.1 or MacDonald criteria for GBM | 4 months
  Tumor responses will be measured according to RECIST 1.1 or MacDonald criteria for GBM

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka

REFERENCES:
- See also: Results for CINC280X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15330